CLINICAL TRIAL: NCT01640171
Title: Topical Lidocaine Gel With and Without Subconjunctival Lidocaine Injection for Intravitreal Injection: a Within-patient Study
Brief Title: Anesthesia Preference for Intravitreal Injection: Topical or Subconjunctival
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Vitreous Associates of Florida (Other)
Responsible Party: Principal Investigator, Steven Cohen, MD, Clinical Professor of Ophthalmology, Retina Vitreous Associates of Florida
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: rvaf-2012
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Age-related Macular Degeneration; Central Retinal Vein Occlusion; Diabetic Macular Edema
Keywords: anesthesia; pain; intravitreal; anti-vegf
MeSH Terms: conditions — Macular Degeneration; Retinal Vein Occlusion; Pain | interventions — Lidocaine; Anesthesia; Anesthetics; proxymetacaine; Tetracaine; Gels; Ketorolac; Anti-Inflammatory Agents; Ranibizumab; Bevacizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Top Anesthesia 1 Eye SC Lidocaine 1 Eye (Other): One eye:
  Proparacaine Hydrochloride 0.5% Drop Tetravisc 0.5% Gel Acuvail Intra-vitreal Anti-VEGF Drug
  Fellow Eye:
  Proparacaine Hydrochloride 0.5% Drop Tetravisc 0.5% Gel Xylocaine 2% Injectable Anesthetic Acuvail Intra-vitreal Anti-VEGF Drug
  Interventions: Procedure: Xylocaine 2% Injectable Anesthetic; Drug: Proparacaine Hydrochloride 0.5% Drop; Drug: Tetravisc 0.5% Gel; Drug: Acuvail; Drug: Intra-vitreal Anti-VEGF Drug

INTERVENTIONS:
Procedure: Xylocaine 2% Injectable Anesthetic — xylocaine 2% injection 0.1 cc
  Other Names: Lidocaine; Subconjunctival; Anesthesia; Anesthetic
Drug: Proparacaine Hydrochloride 0.5% Drop — Topical drop given first to the treated eye.
  Other Names: Lidocaine; Topical; Anesthesia; Anesthetic
Drug: Tetravisc 0.5% Gel — Gel applied to eye 3 times prior to treatment
  Other Names: topical; Anesthesia; Anesthetic
Drug: Acuvail — Anti-inflammatory drop given after treatment
  Other Names: anti-inflammatory; ketorolac; topical
Drug: Intra-vitreal Anti-VEGF Drug — Intravitreal injection treating wet AMD or Diabetic Macular Edema or Retinal Vein Occlusion
  Other Names: Lucentis; Avastin; Eylea

SUMMARY:
Since 2004, intravitreal injection of Avastin, Lucentis, and Macugen for wet age-related macular degeneration, retinal vein occlusion, and diabetic macular edema are being administered in the United States at increasing rates. A 2010 study showed that in Canada and the incidence of injections grew 8 fold from 2005 to 2007 to 25.9 injections per 100,000 citizens. (Campbell 2010) In 2009, in the United States, over 1 million intravitreal injections were administered to Medicare beneficiaries. (Wykoff 2011) In the year 2011, the four doctors in my retina group administered a total of 6,494 intravitreal injections; in 2010, we administered 5021 intravitreal injections.

Even though intravitreal injections are commonly administered, the optimal method of anesthetizing the eye prior to injection has yet to be determined. Some physicians use an anesthetic drop, some a soaked cotton pledget, some use an anesthetic gel and some use subconjunctival injected anesthetic.

In 2009, the last time the Procedures and Trends Survey (PAT) (Mittra 2009) conducted by the American Society of Retina Specialists (the largest retina society in the world) asked about anesthetic methods for administering intravitreal injections, the following response was given by the 433 respondents:

* Topical anesthetic drop: 21.48%
* Topical viscous anesthetic: 23.33%
* Topical anesthetic & soaked cotton-tip or pledget: 29.79%
* Subconjunctival injection of anesthetic: 24.02%
* Other: 1.39%

An editorial in 2011 in the journal Retina, discusses the lack of good studies assessing optimal anesthetic prior to intravitreal injections. (Prenner 2011).

DETAILED DESCRIPTION:
Topical lidocaine gel with and without subconjunctival lidocaine injection for intravitreal injection: a within-patient study

Research Protocol

Steven M. Cohen, MD

1 & 2. General information including the rationale for the study. Explain the area of Current scientific concern and why the research is needed; Background information including a description of existing research and information that is already known on the topic; Since 2004, intravitreal injections of Avastin, Lucentis, and Macugen for wet age-related macular degeneration, retinal vein occlusion, and diabetic macular edema are being administered in the United States at an increasing rate. In Canada, the incidence of intravitreal injections grew 8 fold from 2005 to 2007 to 25.9 injections per 100,000 citizens. (Campbell 2010) In 2009, in the United States, over 1 million intravitreal injections were administered to Medicare beneficiaries. (Wykoff 2011) In the year 2011, the four doctors in my retina group administered a total of 6,494 intravitreal injections; in 2010, we administered 5021 intravitreal injections.

Even though intravitreal injections are commonly administered, the optimal method of anesthetizing the eye prior to injection has yet to be determined. Some physicians use an anesthetic drop, some use a soaked cotton pledget, some use an anesthetic gel and some use subconjunctival injected anesthetic.

In 2009, the last time the Procedures and Trends Survey (PAT) (Mittra 2009) conducted by the American Society of Retina Specialists (the largest retina society in the world) asked about anesthetic methods for administering intravitreal injections, the following response was given by the 433 respondents:

* Topical anesthetic drop: 21.48%
* Topical viscous anesthetic: 23.33%
* Topical anesthetic & soaked cotton-tip or pledget: 29.79%
* Subconjunctival injection of anesthetic: 24.02%
* Other: 1.39%

In 2005, 12 patients were studied who were given subconjunctival lidocaine injection prior to intravitreal injection and subsequently (on another visit) given topical gel anesthesia prior to intravitreal injection. The patients rated their pain on a scale from 0 to 10. These researchers found that the pain scores were the same for the two groups but the patients receiving subconjunctival anesthetic had more chemosis and subconjunctival hemorrhage. This study was very small and not powered to determine a difference between the groups. (Friedman 2005)

In 2006, a study comparing topical gel to subconjunctival lidocaine injection using an analog pain scale in one hundred patients found no difference between the two groups (N=100). The intravitreal injection was given within 30 seconds of the first anesthetic application: the application of anesthetic gel or the injection of subconjunctival lidocaine. (Freeman 2006) In most patients, lidocaine take longer than 30 seconds to work. A study of 2% lidocaine for dental procedures shows that the onset of anesthetic for the tooth is 3.3 +/- 1.5 minutes (average +/- SD).(Oka 1997)

In 2012, a study comparing various topical anesthetic agents was published showing no significant difference between topical proparicaine drops, 4% lidocaine solution, and 3.5% lidocaine gel in a group of 120 patients using an analog pain scale from 0 to 10. This study performed the intravitreal injection from between 20 to 70 seconds of the first anesthetic application. (Davis 2012)

In 2012, a study was performed in 60 patients comparing tetracaine, proparacaine, and TetraVisc gel and found tetracaine to be the least painful. They also found significantly lower pain scores in patients who had improved vision from previous injections, female sex, and age > 65. This suggests that factors other than anesthetic type used might affect the results of pain studies. (Rifkin, 2012)

An editorial in 2011 in the journal Retina, discusses the lack of good studies assessing optimal anesthetic prior to intravitreal injections. (Prenner 2011).

3. The research questions, objectives and purpose;

To determine if topical gel with subconjunctival lidocaine is superior to topical gel in relieving pain of intravitreous injection of anti-vascular endothelial growth factor medication.

4. The study design including information that is needed to answer the research questions;

Study Design: This is a within patient, factorial, single blinded, randomized trial comparing topical anesthetic gel to topical anesthetic gel plus subconjunctival lidocaine for relieving pain of intravitreous injections.

Patients receiving bilateral simultaneous injections for wet macular degeneration or retinal vein occlusion or diabetic macular edema will be asked to participate in the study. Those who consent and sign an approved informed consent will be treated as follows:

A coin will be flipped to determine which treatment the right is going to get. The right eye will always be treated before the left eye, but both eyes will be treated as nearly simultaneously as possible. Both eyes will be prepared simultaneously and the left eye will receive its intravitreal injection within 30 seconds of the right eye being injected.

In preparation for the injection, one drop of Proparicaine Hydrochloride 0.5% and one drop brimonidine 0.2%, will be instilled into each eye followed by ¼ inch of TetraVisc Forte Gel. The patient will then be instructed to close the eyes for 5-minutes. Then another application of ¼ inch of TetraVisc Forte Gel will be placed in the inferior conjunctival fornix. Another 5-minute waiting period will be observed. Finally, in the eye randomized to subconjunctival lidocaine 0.1 cc of 2% lidocaine hydrochloride, 20 mg/ml, will injected subconjunctivally at the intended site of the intravitreal injection. In the eye randomized to no subconjunctival lidocaine, a pretend injection will be given by pushing a syringe without a needle against the eye. Another 5-minute waiting period will be observed.

Another drop of Proparicaine Hydrochloride Solution 0.5% will be placed in each eye and another ¼ inch of TetraVisc Gel, and then a sterile eyelid speculum will be used to separate the lid, and then the eyes will be prepped with a drop of 5% Betadine Solution. After the Betadine prep, each eye (right then left) will be injected through the pars plana, 3 mm posterior to the corneal scleral limbus, with the anti-vascular endothelial growth factor drug. Following the intravitreal injection, the sterile lid speculum will be removed. The eyes will be irrigated with sterile eye rinse eye irrigation solution and a drop of Acuvail will be placed into each eye.

The patient will be asked to keep the eyes mostly closed for one hour following the injection, to use artificial tears hourly for every four hours, and to not rub their eyes after the procedure because of the anesthetic. The patient will also be warned to report any adverse events immediately, especially escalating pain, within a day or two after the procedure.

Pain will be rated in two ways during the procedures, comparing the two eyes and also on a 0 to 10 standardized pain scale.

* Prior to any treatment
* After subconjunctival anesthetic
* After intravitreal injection
* That evening by phone
* The following day by phone

At each of these 5 times, patients will be asked if in the right eye compared to the left eye is there:

* Much more pain right eye; a little more pain right eye; no difference; a little more pain left eye; much more pain left eye.
* Rate pain in each eye from 0 to 10

The final endpoint will be the following day when patients decide which eye they prefer overall anesthetic therapy. They will be asked to choose the method for the next visit to be used in both eyes.

If patients do not have a preference after one study visit, a second study visit will be performed reversing treatment as to which eye gets which anesthesia. Then they will have to choose which method they like best or state the two treatments are the same.

5. Sample size should be justified

A sample size of 44 patients would provide an 80 percent probability of detecting an important difference in pain magnitude if one exists assuming a ratio of expected treatment effect to standard deviation of 0.6 (two-tailed, alpha = 0.05) (Friedman 2006)

9. The risks to the subjects;

These treatments and anesthetics have been validated in several large clinical studies. There are is a higher risk of subconjunctival hemorrhage and chemosis in eyes with a subconjunctival anesthetic. Neither of those causes lasting harm to the eye, but they can cause some discomfort for a day or two. With either anesthetic, there is a risk of: conjunctival hemorrhage, eye pain, vitreous floater, foreign body sensation, and ocular discomfort.

10.Any experimental procedures including the use procedures already being performed on subjects for diagnostic or treatment purposes;

None.

11.The potential benefits to subjects;

This study will allow each patient to determine the optimal anesthetic protocol for themselves. From experience, there are some patients who prefer one mode of anesthesia and some who prefer another mode of anesthesia. Usually the physician chooses the anesthetic type. This study will allow each patient to determine what type of anesthetic they prefer.

12.Human subjects considerations including a description of the informed consent process; when potentially vulnerable subjects will be enrolled (e.g., children, prisoners, the cognitively impaired, institutionalized or critically/terminally ill), include a discussion of additional safeguards in place to protect the subjects; include a discussion of how the privacy and confidentiality of the subjects will be maintained

Informed consent will be given both verbal and written on the day of the visit. Patients who are eligible will also be contact by phone prior to the visit so they can be told about the study on the phone. Finally, patients will be given the option to enter or leave the study whenever they want. If they do not want to enroll on the initial visit when the study is discussed, they will be offered entry on the following visit. No children, prisoners, cognitively impaired or terminally ill patients will be enrolled. Finally, all research notes will only have a code using the patient's record number from our retina practice on it. Charts in our office are always maintained in a HIPPA compliant manner.

13.Data and safety monitoring plan including whether or not there is a data and safety monitoring board associated with the study, how often data will be reviewed for safety, early stopping criteria, etc.

There is no data and safety monitoring board.

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving bilateral intravitreal injections
* Ability to give informed consent

Exclusion Criteria:

* Pre-existing eye pain
* Uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Cohen, MD, Principal Investigator — Retina Vitreous Associates of Florida
Locations (1):
- Retina Vitreous Associates of Florida, Clearwater, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Anesthesia 1 Eye, SC 1 Eye: Eye receiving only topical gel
  Proparacaine Hydrochloride 0.5% Drop: Topical drop given first to the treated eye.
  Tetravisc 0.5% Gel: Gel applied to eye 3 times prior to treatment
  Acuvail: Anti-inflammatory drop given after treatment
  Intra-vitreal Anti-VEGF Drig: Intravitreal injection treating wet AMD or Diabetic Macular Edema or Retinal Vein Occlusion
  Fellow eye Same as above plus Xylocaine 2% SC
Period: Overall Study
Arm/Group | Topical Anesthesia 1 Eye, SC 1 Eye
Started | 57
Completed | 57
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 57 patients were treated differently in each eye.
Groups:
- Topical Anesthesia 1 Eye, SC 1 Eye: Eye receiving only topical gel
  Proparacaine Hydrochloride 0.5% Drop: Topical drop given first to the treated eye.
  Tetravisc 0.5% Gel: Gel applied to eye 3 times prior to treatment
  Acuvail: Anti-inflammatory drop given after treatment
  Intra-vitreal Anti-VEGF Drig: Intravitreal injection treating wet AMD or Diabetic Macular Edema or Retinal Vein Occlusion
  Fellow Eye:
  Eye receiving topical gel and subconjunctival lidocaine
  Xylocaine 2% Injectable Anesthetic: xylocaine 2% injection 0.1 cc
  Proparacaine Hydrochloride 0.5% Drop: Topical drop given first to the treated eye.
  Tetravisc 0.5% Gel: Gel applied to eye 3 times prior to treatment
  Acuvail: Anti-inflammatory drop given after treatment
  Intra-vitreal Anti-VEGF Drig: Intravitreal injection treating wet AMD or Diabetic Macular Edema or Retinal Vein Occlusion
Arm/Group | Topical Anesthesia 1 Eye, SC 1 Eye
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 82 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Preferred Subconjunctival Anesthetic at the Third Follow-up Visit
Description: Participants received anesthetic over several treatment visits. They were allowed to change there preference at each visit. The final outcome was the preference indicated at the third follow-up visit.
Time Frame: up to 6 months
Measure: Number; unit: participants
Groups:
- Topical Anesthesia 1 Eye, SC 1 Eye: Eye receiving only topical gel
  Proparacaine Hydrochloride 0.5% Drop: Topical drop given first to the treated eye.
  Tetravisc 0.5% Gel: Gel applied to eye 3 times prior to treatment at three minute intervals
  Acuvail: Anti-inflammatory drop given after treatment
  Intra-vitreal Anti-VEGF Drig: Intravitreal injection treating wet AMD or Diabetic Macular Edema or Retinal Vein Occlusion
  Fellow eye:
  Same as above plus SC Xylocaine was administered following the first two topical anesthetic applications
Arm/Group | Topical Anesthesia 1 Eye, SC 1 Eye
Number analyzed (Participants) | 57
participants | 50

2. Secondary Outcome: Number of Participatns With Level 10 Pain on Wong-Baker Pain Scale In Subconjunctival Eye At Time of Intravitreal Injection
Description: Pain was rated on a 10 point standardized pain scale, zero was the least pain and 10 was the worst pain. The patient was questioned using a script and shown a pain scale as well as told how the pain scale worked. Then the patient gave the number that characterized their pain.
Time Frame: 24 hours
Population: All patients in the study
Measure: Number; unit: participants
Arm/Group | Topical Anesthesia 1 Eye, SC 1 Eye
Number analyzed (Participants) | 57
participants | 0

3. Secondary Outcome: Likert Like Pain Scale Number of Participants Who Said the Topical Eye Hurt Much More Than the Subconjunctival Eye at Time of Intravitreal Injection
Description: The patient was asked to compare the two eyes in the way described in the study protocol on a five point scale. If one eye hurt a lot more or a little more than the other or if the two eyes were equal (neither hurt more than the other).
Time Frame: 24 hours
Population: total group
Measure: Number; unit: participants
Arm/Group | Topical Anesthesia 1 Eye, SC 1 Eye
Number analyzed (Participants) | 57
participants | 19

ADVERSE EVENTS:
Time Frame: 1 year
Description: Patients were followed for a total of one year
Groups:
- Topical Anesthesia: Eye receiving only topical gel
  Proparacaine Hydrochloride 0.5% Drop: Topical drop given first to the treated eye.
  Tetravisc 0.5% Gel: Gel applied to eye 3 times prior to treatment
  Acuvail: Anti-inflammatory drop given after treatment
  Intra-vitreal Anti-VEGF Drig: Intravitreal injection treating wet AMD or Diabetic Macular Edema or Retinal Vein Occlusion
- Subconjunctival Anesthesia: Eye receiving topical gel and subconjunctival lidocaine
  Xylocaine 2% Injectable Anesthetic: xylocaine 2% injection 0.1 cc
  Proparacaine Hydrochloride 0.5% Drop: Topical drop given first to the treated eye.
  Tetravisc 0.5% Gel: Gel applied to eye 3 times prior to treatment
  Acuvail: Anti-inflammatory drop given after treatment
  Intra-vitreal Anti-VEGF Drig: Intravitreal injection treating wet AMD or Diabetic Macular Edema or Retinal Vein Occlusion
Arm/Group | Topical Anesthesia | Subconjunctival Anesthesia
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 0/57 | 0/57

LIMITATIONS AND CAVEATS:
Most patients were treated with subconjunctival anesthetic prior to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No